CLINICAL TRIAL: NCT04359654
Title: A Single-site, Randomised, Controlled, Parallel Design, Open-label Investigation of an Approved Nebulised Recombinant Human DNase Enzyme (Dornase Alfa) to Reduce Hyperinflammation in Hospitalised Participants With COVID-19
Brief Title: Nebulised Dornase Alfa for Treatment of COVID-19 (Coronavirus Disease 2019)
Acronym: COVASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132333
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: COVID-19 (Coronavirus Disease 2019); Hypoxia
Keywords: COVID; COVID19; Pneumonia; Coronavirus; Hypoxia; C-Reactive Protein
MeSH Terms: conditions — COVID-19; Hypoxia; Pneumonia; Coronavirus Infections | interventions — dornase alfa

STUDY DESIGN:
Intervention Model Description: An open-label, randomised, Best-Available-Care (BAC) and historic-controlled trial of nebulised dornase alfa [2.5 mg BID] for 7 days in participants with COVID-19 who are admitted to hospital and are at risk of ventilatory failure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dornase alfa treatment (Experimental): Best available care and nebulised dornase alfa [2.5 mg BID] for 7 days in participants with COVID-19 who are admitted to hospital and are at risk of ventilatory failure
  Interventions: Drug: Dornase Alfa Inhalation Solution [Pulmozyme]
- Best available care (No Intervention): Best available standard of care

INTERVENTIONS:
Drug: Dornase Alfa Inhalation Solution [Pulmozyme] — Nebulised Dornase alfa 2.5mg bd for 7 days
  Arms: Dornase alfa treatment

SUMMARY:
An open-label, randomised, Best-Available-Care (BAC) and historic-controlled trial of nebulised dornase alfa [2.5 mg BID (bis in die)] for 7 days in participants with COVID-19 who are admitted to hospital and are at risk of ventilatory failure (the COVASE study). Controls will include a randomised arm to receive BAC, historic data from University College London Hospitals NHS Foundation Trust (UCLH) patients with COVID-19 and biobanked samples will be used to demonstrate an effect of dornase alfa. C-reactive protein (CRP) will be measured to assess the effect of dornase alfa on inflammation. Clinical endpoints and biomarkers (e.g. d-dimer) will be used to assess the clinical response. Exploratory endpoints will explore the effects of dornase alfa on features of neutrophil extracellular traps (NETs).

DETAILED DESCRIPTION:
Dornase alfa is a recombinant human DNase enzyme indicated in conjunction with standard therapies for the management of cystic fibrosis (CF) to improve pulmonary function. Dornase alfa degrades extracellular DNA, and so promotes the clearance of NETs and lead to a significant improvement in lung function for treated CF patients by facilitating mucus clearance in the lung. Dornase alfa is approved worldwide as a nebulised formulation, with an excellent safety profile and is well tolerated. The most common side effect is a hoarse voice. Moreover, dornase alfa could be administered in addition to effective antiviral therapy and should not interfere with antiviral drugs that could be used for COVID-19.

By facilitating the clearance of NETs, dornase alfa not only facilitates sputum clearance in CF patients, but has additional anti-inflammatory activity. Dornase alfa has been shown to reduce NETs in the bronchoalveolar lavage (BAL) and sputum of participants with CF (Konstan et al 2012). In the Bronchoalveolar Lavage for the Evaluation of Anti-inflammatory Treatment (BEAT) study, the percentage of neutrophils in bronchoalveolar lavage fluid significantly increased in untreated CF patients (P<0.02) while remaining constant in the dornase alfa-treated group. Levels of elastase and IL-8 also significantly increased from baseline in the untreated group (P<0.007 and P<0.02 for elastase and IL-8, respectively), but remained stable in patients receiving dornase alfa (Konstan and Ratjen, J. Cyst. Fibros. 2012).

There is scientific evidence to support the potential benefits of dornase alfa in COVID-19 infection. Viral sepsis driven by a hyperinflammation is thought to be a major cause of mortality in COVID-19 infection. Interleukin-1β (IL-1β), IL-6 and TNFα (tumour necrosis factor alpha) are key cytokines in microbial sepsis. Positive outcomes with Roche's Actemra (tocilizumab), an antibody that blocks the pro-inflammatory cytokine interleukin-6 (IL-6), in COVID-19 treatment has led to several anti-inflammatory trials.

Our hypothesis is that nebulised dornase alfa will break down the DNA backbone of NETs in the COVID-19 lung which will promote the degradation of pro-inflammatory extracellular histones and prevent the amplification of the inflammatory response and the resultant lung damage.

Positive data will enable rapid testing into a large clinical trial in the UK (United Kingdom) and prevent ICU (intensive care unit) capacity issues faced today. Dornase alfa is a cost-effective drug and is currently available for prescription.

We propose to test this hypothesis with this COVASE Phase 2a trial. We propose that all people with COVID-19 who are admitted to hospital for supplementary oxygen, who showed evidence of systemic inflammation but did not immediately require intubation and ventilation, would be eligible for nebulised Dornase alfa, a safe and cost-effective treatment, twice daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants, aged ≥ 18 years.
2. Participants who are hospitalised for suspected Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test or radiological confirmation.
3. Participants with stable oxygen saturation (>=94%) on supplementary oxygen
4. CRP >= 30 mg/L.
5. Participants will have given their written informed consent to participate in the study and are able to comply with instructions and nebuliser.

Exclusion Criteria:

1. Females who are pregnant, planning pregnancy or breastfeeding.
2. Concurrent and/or recent involvement in other research or use of another experimental investigational medicinal product that is likely to interfere with the study medication within the last 3 months before study enrolment.
3. Serious condition meeting one of the following:

   I. respiratory distress with respiratory rate >=40 breaths/min II. oxygen saturation <=93% on high-flow oxygen
4. Require mechanical invasive or non-invasive ventilation at screening
5. Concurrent severe respiratory disease such as asthma, COPD (chronic obstructive pulmonary disease) and/or ILD (interstitial lung disease).
6. Any major disorder that in the opinion of the Investigator would interfere with the evaluation of the results or constitute a health risk for the study participant.
7. Terminal disease and life expectancy <12 months without COVID-19.
8. Known allergies to the dornase alfa and excipients.
9. Participants who are unable to inhale or exhale orally throughout the entire nebulisation period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Porter, MD PhD, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised results will be published in a scientific journal (TBC) and posted on the Breathing Matters website www.breathingatters@ucl.ac.uk

REFERENCES:
- [Derived] Porter JC, Inshaw J, Solis VJ, Denneny E, Evans R, Temkin MI, De Vasconcelos N, Aramburu IV, Hoving D, Basire D, Crissell T, Guinto J, Webb A, Esmail H, Johnston V, Last A, Rampling T, Lippert L, Helbig ET, Kurth F, Williams B, Flynn A, Lukey PT, Birault V, Papayannopoulos V. Anti-inflammatory therapy with nebulized dornase alfa for severe COVID-19 pneumonia: a randomized unblinded trial. Elife. 2024 Jul 16;12:RP87030. doi: 10.7554/eLife.87030. PMID 39009040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from acute COVID-19 (Coronavirus Disease 2019) wards between between May 2020-October 2021
Groups:
- Dornase Alfa Treatment: Best available care and nebulised Dornase alfa [2.5 mg BID (bis in die)] for 7 days in participants with COVID-19 who are admitted to hospital and are at risk of ventilatory failure
  Dornase alfa Inhalation Solution [Pulmozyme]: Nebulised Dornase alfa 2.5mg bd for 7 days
Period: Overall Study
Arm/Group | Dornase Alfa Treatment | Best Available Care
Started | 31 | 10
Completed | 30 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dornase Alfa Treatment | Best Available Care | Total
Number analyzed (Participants) | 30 | 9 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (12.5) | 53.3 (13.7) | 56.8 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 23 | 7 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
C-reactive protein [Mean (Standard Deviation); unit: mg/L] — mg/L Serum measurement
  mg/L | 101.9 (52.2) | 91.9 (68.1) | 100.2 (63.3)
Co-morbidities [Count of Participants; unit: Participants] | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Measuring the Change in Inflammation
Description: Analysing stabilisation of C-reactive protein.
Time Frame: 7 days
Population: The reported LS (least squares) means are antilogs of the LS means estimated on the log scale.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/L
Groups:
- Best Available Care (Randomised): Best available standard of care of patients randomised (9)
Arm/Group | Dornase Alfa Treatment | Best Available Care (Randomised)
Number analyzed (Participants) | 30 | 9
mg/L | 23.23 [17.71 to 30.46] | 34.82 [28.55 to 42.47]
Statistical Analysis 1: Comparison: Dornase Alfa Treatment vs Best Available Care (Randomised); Test type: Superiority; p = 0.01, Mixed Models Analysis

2. Secondary Outcome: Survival at 35 Days
Description: Survival at 35 days (28 days post last treatment day) Participants were followed up until discharge or death or a maximum of 28 days post last treatment day.
Time Frame: 35 days
Population: Patients alive at 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dornase Alfa Treatment | Best Available Care (Randomised)
Number analyzed (Participants) | 30 | 9
Participants | 29 | 9
Statistical Analysis 1: Comparison: Dornase Alfa Treatment vs Best Available Care (Randomised); Test type: Superiority; p = 0.03, Mixed Models Analysis

3. Secondary Outcome: Discharge Before 35 Days
Description: Number of participants discharged before 35 days
Time Frame: Before 35 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dornase Alfa Treatment | Best Available Care
Number analyzed (Participants) | 30 | 9
Participants | 27 | 8

4. Secondary Outcome: D-dimer (ug/L)
Description: Change in D-dimer (ug/L) The reported LS means are antilogs of the LS means estimated on the log scale.
Time Frame: 7 days
Population: Those that had d-dimer measured.
Measure: Least Squares Mean (95% Confidence Interval); unit: (ug/L) FEU
Arm/Group | Dornase Alfa Treatment | Best Available Care (Randomised)
Number analyzed (Participants) | 28 | 9
(ug/L) FEU | 570.78 [384.51 to 847.3] | 1656.96 [876.93 to 3130.81]
Statistical Analysis 1: Comparison: Dornase Alfa Treatment vs Best Available Care (Randomised); Test type: Superiority; p = 0.004, Mixed Models Analysis

5. Secondary Outcome: Lymphocyte Count (×109/L)
Description: measure of Lymphocyte count (×109/L)
Time Frame: 7 days
Population: The reported LS means are antilogs of the LS means estimated on the log scale.
Measure: Least Squares Mean (95% Confidence Interval); unit: ×10^9 cells/L
Arm/Group | Dornase Alfa Treatment | Best Available Care (Randomised)
Number analyzed (Participants) | 30 | 9
×10^9 cells/L | 1.08 [0.92 to 1.27] | 0.87 [0.76 to 0.98]
Statistical Analysis 1: Comparison: Dornase Alfa Treatment vs Best Available Care (Randomised); The reported LS means are antilogs of the LS means estimated on the log scale; Test type: Superiority; p = 0.021, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 35 days or discharge whichever was sooner
Groups:
- Dornase Alfa Treatment: Best available care and nebulised dornase alfa [2.5 mg BID] for 7 days in participants with COVID-19 who are admitted to hospital and are at risk of ventilatory failure
  Dornase Alfa Inhalation Solution [Pulmozyme]: Nebulised Dornase alfa 2.5mg bd for 7 days
  Note: Adverse events for matched historic controls were not recorded.
  Participants were followed up until discharge or death or a maximum of 28 days post last treatment day.
- Best Available Care: Best available standard of care Note: Adverse events for matched historic controls were not recorded. Participants were followed up until discharge or death or a maximum of 28 days post last treatment day.
Arm/Group | Dornase Alfa Treatment | Best Available Care
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/9
Serious Adverse Events (participants affected / at risk) | 8/30 | 2/9
Other Adverse Events (participants affected / at risk) | 16/30 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dornase Alfa Treatment (N=30) | Best Available Care (N=9)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure type 2 (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure type 1 (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Aspiration pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Hospital acquired pneumonia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dornase Alfa Treatment (N=30) | Best Available Care (N=9)
Chest pain (General disorders) | 3 (3) | 0 (0)
Chest tightness (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum bloody (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Confusion aggravated (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disturbance (Psychiatric disorders) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Cognitive impairment (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizzy spells (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Tingling feet/hands (Nervous system disorders) | 1 (1) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tingling mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcerative colitis relapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Transaminitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Leg spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-04-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT04359654/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04359654/SAP_001.pdf